CLINICAL TRIAL: NCT04991701
Title: The Natural History of Ataxia Telangiectasia
Brief Title: A National Retrospective Population Based Cohort Study of the Natural History of Ataxia Telangiectasia
Acronym: N-HAT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); Royal Papworth Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 16069
Record Dates: First submitted 2021-06-30; First posted 2021-08-05 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Ataxia Telangiectasia
Keywords: Ataxia; Telangiectasia; Epidemiology
MeSH Terms: conditions — Ataxia Telangiectasia; Ataxia; Telangiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective observational study of natural-history of ataxia-telangiectasia. Understanding the natural history and its variability is not only vital to planning effective patient-centred services, and counselling patients and their families, but will also inform the design of future clinical research, particularly clinical trials.

DETAILED DESCRIPTION:
Ataxia Telangiectasia (A-T), a life shortening autosomal recessive multisystem disease, is caused by mutations in the ATM gene, and affects 1/300,000 live births. The pathophysiological basis of the disease relates to mutations in the ATM kinase gene that result in a faulty repair of breakages in double-stranded DNA. A-T causes a progressive ataxia, dystonia, and movement disorder, and is complicated by immunodeficiency, lung disease, faltering growth, limb and spinal deformities, and increased susceptibility to cancers. The disease first manifests in early childhood with balance problems and is slowly progressive, with loss of control of limb and eye movements, and speech, through the school years, resulting in severe disability by adulthood. Patients with classical A-T rarely live beyond their 20s, and there is no effective treatment. Because it is so rare, little has been published on the natural history of the condition.

The Department of Health funds the national multidisciplinary clinic for children with A-T in Nottingham, with follow-up of adults at the Royal Papworth Hospital, Cambridgeshire. Clinical and laboratory data have been collected systematically from over 170 patients, most on more than one occasion, from 2001 to date. This unique clinical collection will allow us to elucidate the natural history of A-T using a mixture of cross-sectional and longitudinal analyses, from presentation in the pre-school years to adulthood.

We will discover more about the presentation and diagnosis of A-T, and the detailed evolution of the disease as children grow to adulthood. Preliminary analyses of the neurological phenotype in 134 patients has shown important genotype-phenotype relationships and a more variable deterioration over time than anticipated, which will be investigated further. In parallel, investigation of the morbidity and mortality due to deterioration in lung function, the immune system, infections, cancers, malnutrition, and skeletal deformity will be undertaken. We will learn about the interactions between the various disease manifestations, e.g. lung disease and nutritional status, immunological impairment and neurology and risk of cancers. These discoveries will inform patient care, and help to generate hypotheses for further research projects. From the analysis of the cross-sectional data we will establish an initial Core Outcome Set, which will be further developed at Patient and Public Involvement (PPI) meetings with young people with A-T and their parents/carers.

This study is needed to accurately map the course of A-T from childhood to adulthood, to help us recognise different patterns of disease in individual patients, improve early diagnosis by understanding the reasons for diagnostic delay, anticipate complications more accurately and elucidate the best ages to intervene before rapid deterioration.

The expected clinical course involves deterioration in gross and fine motor skills, oculomotorpraxia, choreoform movements, and difficulty with chewing and swallowing. By the end of their first decade children are usually wheelchair dependent as cerebellar destruction progresses and further neurodisability ensues with development of incapacitating movement disorder and peripheral neuropathy. Sinopulmonary infections and recurrent lower respiratory tract infections with bronchiectasis are common in A-T, and current management aims to avoid and treat lung infection. The treatment for malignancy must take into consideration the fact that many oncological therapies have adverse-effects that will impact on individual function in other domains for example drugs that cause muscle weakness will exacerbate motor impairments. Also the DNA of patients with A-T is particularly susceptible to double strand breakage, which can itself cause secondary malignancies.

Understanding the natural history and its variability is not only vital to planning effective patient-centred services, and counselling patients and their families, but will also inform the design of future clinical research, particularly clinical trials. The choice of age group to include in a trial, duration of treatment, and choice of core outcome measures will depend on the results of this natural history study.

This study will centre on data analysis and will not involve any therapeutic interventions, although it is intended that the results will enable future research to determine optimum therapeutic strategies. The benefits of this study thus relate to the compilation of vast amounts of data that have been gathered on A-T over the last 15 years and extracting meaningful information that will inform future care. There is no identifiable risk from inclusion in the study as it involves patient data that are gathered through standard clinical interaction and does not involve introducing or changing treatments or any increased patient interaction apart from voluntary participation of a sample of parents / guardians and young people with A-T in the PPI focus group meetings, for which informed consent will be sought.

There are no established treatments for A-T. Symptomatic treatments are used in patients depending on their symptoms, e.g. gastrostomy feeds are used when eating becomes too slow, or too difficult because of swallowing difficulties. Antibiotics and chest physiotherapy are used to prevent and treat chest infections. Immunodeficiency can be treated in selected cases, as can the various complications of A-T as and when they arise, including scoliosis, cancers, granulomas, movement disorders and spasticity.

Current therapy in A-T is aimed at mitigating neurological deterioration, prevention and treatment of respiratory complications, early identification and treatment of malignancy whilst minimising adverse-effects and treating immunodeficiency with immunoglobulin, in other words, managing the downstream complications of the gene mutation. Each aspect and complication requires specialist assessment and input and monitoring of progression and response to treatment. A-T is managed from a multi-speciality and multi-disciplinary perspective and in Nottingham this happens in the setting of the National A-T Clinic that children attend with their families every two years. Neurological progression is determined using the A-T Index and AT-NEST scoring systems. Assessment by a clinician with paediatric respiratory expertise also occurs alongside input from a neurologist, immunologist, geneticist, dietician, occupational and physiotherapist, clinical psychologist and speech and language therapist. One of the aims of this natural history study is to avoid complications developing by elucidating the optimal timing of treatment interventions.

Respiratory disease patterns in A-T include sinopulmonary disease and bronchiectasis, interstitial lung disease and lung disease associated with neuromuscular, especially bulbar, dysfunction. At present treatment depends on the pattern of lung disease and can range from antibiotics, immunoglobulin replacement, systemic steroids, chest physiotherapy, and steps to limit aspiration. Assessment of response to treatment includes assessment of resolution or persistence of symptoms, spirometry measurements, and imaging such as chest x-rays and where indicated, CT scans, although limiting exposure to radiation is always a factor to consider in patients with A-T.

There have been several small scale pilot trials of medication for the neurological impairments with mixed success, including the use of amantidine5, betamethasone6,7, and dexamethasone loaded autologous redcells8.

Potential but as yet untested treatments include anti-oxidants which have the potential to slow down progression of neurodegeneration by protecting Purkinje cells in the cerebellum from oxidative stress caused by free radicals. ATM has a role in the inhibition of oxidative stress and absence or reduced function of ATM could result in increased oxidative stress and accelerated neuronal loss.11

However, all these suggestions in fact impact the downstream consequences of the mutations. In cystic fibrosis, another multisystem genetic disease which largely impacts the respiratory system, the treatment paradigm has shifted from downstream treatment of the consequences of gene dysfunction, to gene therapy and small molecule treatments addressing the basic defect. It is likely that in the near future A-T will follow this paradigm, e.g. with the development of drugs to allow read-through of premature termination codons, or the skipping of mutations, or the incorporation of functioning genetic sequences into the genome. These and other, as yet unknown, therapeutic approaches will require carefully designed clinical trials, and this natural history study will inform the design of such future trials.

The study will allow a systematic approach to A-T and an understanding of the progression of respiratory, neurological, immunological and oncological disease that underline this multi-systemic disorder, as well as the impact of growth impairment. It will enable evaluation of procedures and medical treatments as well as surgical therapies. There will be insight into the psychological impact of the illness of children and their families and whether there is a particular period where increased or additional support needs to be offered.

As discussed earlier, a critical outcome will be determining the timing of appropriate therapeutic interventions to prevent complications and delay progression of disease, as well as the potential to inform the design of future clinical trials involving therapies for A-T. As a natural history study there will be scope to extract information about A-T within all domains and identify any important variables in treatment, identify whether timing of treatment needs adjustment for maximal impact, for example, by earlier introduction of therapy there may be slower progression of disease or fewer complications.

A possible negative consequence is that the information gleaned might be of little immediate clinical use, however we do not think that will be the case. We think that the data will be valuable in highlighting evidence gaps and informing new studies. We may find that there are inconsistencies in treatments offered to patients and which will encourage us to try to rationalise and streamline our clinical assessments and advice.

ELIGIBILITY:
Inclusion Criteria:

* All patients, with a clinical diagnosis of A-T who have attended the UK's National Ataxia-Telangiectasia clinic in Nottingham or the national adult A-T service in Papworth, of any age

Exclusion Criteria:

* Patients aged 16 and over who specifically inform us that they do not want their clinical data included in the study.
* Patients aged under 16 whose parents / guardian inform us that they do not want their child's clinical data included in the study.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The UK Department of Health funds the national multidisciplinary clinic for children with A-T in Nottingham, with follow-up of adults at the Royal Papworth Hospital, Cambridgeshire. These clinics cover the whole NHS service in the UK and is the tertiary referral clinic or all cases in the country.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Age at diagnosis | through study completion, an average of 1 year
  Age (in months) at which a formal diagnosis of A-T was given
Age of death | through study completion, an average of 1 year
  Age of death of patient with diagnosis of A-T

SECONDARY OUTCOMES:
Age at onset of ataxia | through study completion, an average of 1 year
  Age at which ataxia was reported for the first time
Age at wheelchair dependence | through study completion, an average of 1 year
  Age at which patient became unable to ambulate without a wheelchair

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Ojha, PhD, Principal Investigator — University of Nottingham
Locations (2):
- United Kingdom (2):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: No